CLINICAL TRIAL: NCT07208019
Title: Study on the Key Technology of Acupoint Modulation-based Brain Electric Field Therapy for the Treatment of Post-stroke Cognitive Impairment
Brief Title: Electroacupuncture Treatment for Post-stroke Cognitive Impairment
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ruijie Ma (Other)
Collaborators: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other); The Third Affiliated hospital of Zhejiang Chinese Medical University (Other); The First Affiliated Hospital of Zhejiang Chinese Medical University (Other); Hangzhou Hospital of Traditional Chinese Medicine (Other); Zhejiang Provincial People's Hospital (Other)
Responsible Party: Sponsor-Investigator, Ruijie Ma, Project sponsor, principal investigator, project leader, professor, The Third Affiliated hospital of Zhejiang Chinese Medical University
Organization: The Third Affiliated hospital of Zhejiang Chinese Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2025C02200
Record Dates: First submitted 2025-09-09; First posted 2025-10-06 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-09

CONDITIONS: Post-Stroke Cognitive Impairment (PSCI)
Keywords: Stroke; PSCI; Post-stroke cognitive impairment
MeSH Terms: conditions — Stroke | interventions — Acupuncture Therapy; Electroacupuncture

STUDY DESIGN:
Who Masked: Participant
Masking Description: In the whole research process the principle of three separations was implemented: the three parties of operators efficacy evaluators and statistical analysts were separated and the three parties could not exchange research data implementation and other related contents during the whole process of the study. That is to say the third-party professional statisticians who did not know the grouping situation carried out the efficacy evaluation and statistical analysis of the result data in order to try to avoid the bias of the data results caused by single blinding.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sham electroacupuncture group (Sham Comparator): Treatment of electroacupuncture device without output current based on ordinary acupuncture and moxibustion
  Interventions: Other: Acupuncture
- Electroacupuncture group (Experimental): Treatment with electro-acupuncture device on the basis of ordinary needling
  Interventions: Other: Acupuncture

INTERVENTIONS:
Other: Acupuncture — Electroacupuncture group: After local routine disinfection.Select the main acupoints of bilateral frontoparietal line (MS2), Tianzhu (BL10), Fengchi (GB20), blood supply, parietal midline (MS5), and parietal midline (MS8). Connect the wires of the electroacupuncture instrument to the same side of the bilateral frontoparietal line(MS2) and Tianzhu acupoint (BL10), and perform head electroacupuncture treatment on both sides with a pair on each side.There are two groups of electroacupuncture, with a continuous frequency of 100Hz, and each electroacupuncture stimulation lasts for 30 minutes. After enrollment, treatment will be conducted 5 times a week for 8 weeks.
  Other Names: Electroacupuncture
  Arms: Electroacupuncture group
Other: Acupuncture — Sham electroacupuncture group: After local routine disinfection. Choose the same acupoints as the electroacupuncture group, but use a specially designed electroacupuncture instrument that cannot output current, with only indicator lights or parameter displays when in use.
  Other Names: Sham electroacupuncture
  Arms: Sham electroacupuncture group

SUMMARY:
Stroke is a global public health issue, and it has become a leading cause of death and disability in China. With the rapid aging of the Chinese population, its incidence rate is continuously rising. According to the "China Stroke Prevention and Treatment Report (2023)", on average, one person experiences a new or recurrent stroke every 10 seconds in China, and one person dies from stroke every 28 seconds. Currently, there are 4 million new stroke cases in China each year, with 12.42 million individuals aged 40 and above currently suffering from stroke, and the affected population is showing a trend of younger onset. Among survivors, approximately 75% suffer from residual disabilities, and 40% have severe disabilities. Consequently, patient families will experience significant economic losses and physical and psychological pain.

Post-Stroke Cognitive Impairment (PSCI) is a common complication of stroke, where patients develop cognitive impairment within six months after the stroke event that meets the diagnostic criteria for cognitive impairment. PSCI is defined as a clinical phenomenon secondary to stroke events, with cognitive decline as its core characteristic. Such impairments encompass cognitive dysfunction caused by various stroke types and are one of the main determinants of functional dependency in post-stroke survivors. The prevalence of PSCI within six months is approximately 30% to 50%, with 10% progressing to dementia. Additionally, PSCI patients face a high risk of death, with up to 61% dying within five years. Countries worldwide have launched targeted guidelines, calling for increased attention and investment in this major complication. However, current treatments for PSCI are still limited to secondary prevention measures for stroke and drugs for treating Alzheimer's disease-like conditions, all lacking high-level clinical evidence. Therefore, effective treatments are urgently needed to improve patient outcomes.

PSCI is a dynamically evolving process, with individual differences in its occurrence time, influencing factors, clinical manifestations, and recovery prognosis. The unique diagnostic system of traditional Chinese medicine may assist in analyzing the disease progression of PSCI. The study of the patterns of syndrome evolution can help explain and provide reference for treatment. Currently, there are no specific drugs for treating PSCI, and relevant drug treatments lack high-level evidence. In recent years, with the development of imaging, artificial intelligence, and electromagnetic physics, non-pharmacological therapies have gradually become one of the research hotspots in the field of PSCI. It is worth noting that non-invasive brain stimulation, represented by transcranial electrical stimulation, is a therapy that directly acts on the brain lesions of PSCI and is often used in combination with acupoint stimulation to achieve better therapeutic effects. Meanwhile, acupuncture and moxibustion therapy has demonstrated good efficacy and safety in the prevention and treatment of PSCI. Multiple clinical studies suggest that electroacupuncture therapy can improve cognitive impairment in patients with PSCI and enhance their quality of life. Furthermore, electroacupuncture therapy can also provide targeted treatment for patients through syndrome differentiation and treatment, compensating for the limitations of Western medicine drug therapy.

This study aims to investigate the evolution patterns of syndromes in post-stroke cognitive impairment (PSCI). Simultaneously, through the standardization of multidimensional and multimodal data related to PSCI patients, we will conduct a multicenter, large-sample clinical randomized controlled trial of electroacupuncture intervention for PSCI using a multimodal artificial intelligence big data model. The goal is to establish a characteristic technology for the diagnosis and treatment of PSCI in traditional Chinese medicine (TCM) that is suitable for promotion, and to establish clinical diagnosis and treatment pathways and standard specifications for diseases where TCM has advantages. This will facilitate the establishment of an efficacy evaluation system for PSCI based on TCM syndrome diagnosis and evolution patterns, realize a precise diagnosis and treatment model combining traditional Chinese and Western medicine for PSCI, and improve patients' overall efficacy and quality of life.

ELIGIBILITY:
Inclusion criteria

* According to the Western diagnostic criteria for vascular cognitive impairment outlined in the "Chinese Guidelines for the Diagnosis and Treatment of Vascular Cognitive Impairment (2024 Edition)" developed by the Vascular Cognitive Impairment Branch of the Chinese Stroke Society.
* Meets the traditional Chinese medicine diagnostic criteria for vascular cognitive impairment in the "Guidelines for Traditional Chinese Medicine Diagnosis and Treatment of Vascular Mild Cognitive Impairment (2024)";
* The Mini Mental State Examination (MMSE) score ranges from 12-24, while the Montreal Cognitive Assessment (MoCA) score is below 24; Having cognitive impairment but not reaching the level of severe dementia; The National Institutes of Health Stroke Scale (NIHSS) score is ≤ 8 points; The Early Dementia Screening Scale (Ascertain Dementia 8, AD-8) score is less than 2 points;
* Age between 35-80 years old;
* Have basic communication skills, with Mandarin as the main language (communication language is sufficient), and have at least one stable caregiver;
* Sign the informed consent form.

Exclusion criteria

* Merge serious primary chronic diseases such as heart, liver, kidney, endocrine system, and hematopoietic system, as well as severe cardiovascular and cerebrovascular diseases;
* Skin diseases or scar constitution such as herpes and ulceration are easy to appear on the body surface, which is not suitable for acupuncture and moxibustion treatment;
* Not suitable for repetitive MRI examinations, such as claustrophobia, arterial aneurysm embolization, etc;
* Patients with cognitive impairment or other severe neurological or mental disorders prior to the onset of this illness, and unstable control;
* Patients identified by other clinical trial personnel as unsuitable for this study;
* Participated in clinical research on related diseases in the past 3 months;

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 340 (Estimated)
Dates: Start 2025-10-05 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-03-30 (Estimated)

PRIMARY OUTCOMES:
Neuropsychological Test Battery(NTB) | Week 0 before treatment, Week 12 after treatment, Week 24 after treatment
Montreal Cognitive Assessment | Week 0 before treatment, Week 12 after treatment, Week 24 after treatment
Mini-Mental State Examination | Week 0 before treatment, Week 12 after treatment, Week 24 after treatment

SECONDARY OUTCOMES:
Modified Barthel Index | Week 0 before treatment, Week 12 after treatment, Week 24 after treatment
Hamilton Depression Scale(HAMD) | Week 0 before treatment, Week 12 after treatment, Week 24 after treatment
  <7 indicates no, 7-17 indicates possible, 17-24 indicates certain,>24 indicates severe depression. The lowest score is 0, and the highest score is 46. The higher the score, the more severe the patient's depression.
Electroencephalogram(EEG) | Pre-treatment, 8th week post-treatment
  Evaluate the quantitative electroencephalogram parameters alpha wave, beta wave, delta wave, and theta wave absolute power, as well as the (delta+theta)/(alpha+beta) ratio (DTABR) and delta/alpha power ratio (DAR), and analyze the correlation between various parameters and cognitive function.
Near-infrared spectroscopy | Pre-treatment, 8th week post-treatment
Modified Rankin Scale(mRS) | Week 0 before treatment, Week 12 after treatment, Week 24 after treatment
  The scoring criteria are 0-5 points, with 0 being completely asymptomatic and 5 being severely disabled.
Pittsburgh sleep quality index(PSQI) | Week 0 before treatment, Week 12 after treatment, Week 24 after treatment
  It consists of seven dimensions: subjective sleep quality, falling asleep time, sleep duration, sleep disturbances, use of hypnotic drugs, daytime functional disorders, and sleep efficiency. Each dimension scores 0-3 points, with a minimum score of 0 and a maximum score of 21 points. The higher the score, the more severe the sleep problem. The total score of the seven dimensions is the PSQI score.
Magnetic Resonance Imaging | Pre-treatment, 8th week post-treatment
Short Form 12 Health Survey(SF-12) | Week 8 after treatment
  This scale covers eight aspects: physical function, physical role, pain, general health, mental health, social function, emotional role, and psychological health. The overall score range is 0-100 points, with higher scores indicating better health conditions.

CONTACTS AND LOCATIONS:
Overall Officials: Ruijie Ma, Principal Investigator — The Third Affiliated hospital of Zhejiang Chinese Medical University
Locations (5):
- China (5):
  - Zhejiang Provincial Hospital of Traditional Chinese Medicine, Hangzhou, Zhejiang
  - Hangzhou Hospital of Traditional Chinese Medicine, Hangzhou, Zhejiang
  - The Second Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - The Third Affiliated Hospital of Zhejiang Chinese Medical University, Hangzhou, Zhejiang
  - Zhejiang Provincial People's Hospital, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: Undecided
When all research plans are completed and all participants have completed the clinical study, data access can be opened.

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-12-10): https://cdn.clinicaltrials.gov/large-docs/19/NCT07208019/Prot_SAP_002.pdf
  • Informed Consent Form (2025-05-25): https://cdn.clinicaltrials.gov/large-docs/19/NCT07208019/ICF_001.pdf